CLINICAL TRIAL: NCT02371122
Title: Spinal Cord Stimulation (SCS) Therapy Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1673
Record Dates: First submitted 2015-02-19; First posted 2015-02-25 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Failed Back Surgery Syndrome; Degenerative Disk Disease; Epidural Fibrosis; Arachnoiditis; Radiculopathies
MeSH Terms: conditions — Failed Back Surgery Syndrome; Arachnoiditis; Radiculopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- RestoreSensor or RestoreUltra Setting 1 (Active Comparator): Therapy Setting 1
  Interventions: Device: Therapy Setting 1 (Medtronic)
- RestoreSensor or RestoreUltra Setting 2 (Active Comparator): Therapy Setting 2
  Interventions: Device: Therapy Setting 2 (Medtronic)
- RestoreSensor or RestoreUltra Setting 3 (Active Comparator): Therapy Setting 3
  Interventions: Device: Therapy Setting 3 (Medtronic)
- RestoreSensor or RestoreUltra Setting 4 (Sham Comparator): Therapy Setting 4
  Interventions: Device: Therapy Setting 4 (Medtronic)

INTERVENTIONS:
Device: Therapy Setting 1 (Medtronic) — RestoreSensor or RestoreUltra Setting 1
  Arms: RestoreSensor or RestoreUltra Setting 1
Device: Therapy Setting 2 (Medtronic) — Medtronic RestoreSensor or RestoreUltra Setting 2
  Arms: RestoreSensor or RestoreUltra Setting 2
Device: Therapy Setting 3 (Medtronic) — Medtronic RestoreSensor or RestoreUltra Setting 3
  Arms: RestoreSensor or RestoreUltra Setting 3
Device: Therapy Setting 4 (Medtronic) — Medtronic RestoreSensor or RestoreUltra Setting 4
  Arms: RestoreSensor or RestoreUltra Setting 4

SUMMARY:
The purpose of this study is to evaluate the effect of different spinal cord stimulation settings in the treatment of leg pain. Subjects will receive a randomized order of four different programmed stimulation settings for 3 weeks each followed by a fifth and final setting.

ELIGIBILITY:
Inclusion Criteria:

* At least 22 years of age or older at the time of informed consent
* Implanted with a Medtronic RestoreSensor or RestoreUltra SCS system for an on-label indication at least 6 months for the treatment of chronic leg pain, with or without back pain
* Implanted with one or more Medtronic leads located in the epidural space within the thoracic area
* Receiving some level of pain relief with current SCS therapy
* On a stable dose (no new, discontinued or changes in) of all prescription pain medications and willing to maintain or only decrease the dose of all prescribed pain medications
* Read and understand English without assistance
* Willing and able to comply with all study procedures, study visits, and be available for the duration of the study

Exclusion Criteria:

* Diagnosed with complex regional pain syndrome (CRPS), peripheral causalgia, or reflex sympathetic dystrophy (RSD), or causalgia
* Has leg, knee, or foot pain unrelated to on-label indication for SCS therapy (for eg, arthritis, knee surgery, etc.)
* Implanted with both a surgical and percutaneous lead
* Implanted with a peripheral lead for subcutaneous or peripheral nerve stimulation
* Has had any of the following procedures:

  * Neuroablative procedure within six months
  * Neurolytic block within two months
  * Injection therapy for pain within four weeks
  * Sympathetic block within two weeks
* Has an active implanted device (besides RestoreUltra or RestoreSensor neurostimulator), whether turned ON or OFF
* Pregnant or lactating, inadequate birth control, or at risk of pregnancy during this study
* Has an untreated psychiatric comorbidity
* Has serious drug-related behavioral issues
* Has active malignancy or has been diagnosed with cancer and has not been in remission for at least one year
* Has secondary gains which, in the opinion of the investigator, are likely to interfere with the study
* Participating or planning to participate in another clinical trial while enrolled in this study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2016-11 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale - Leg pain | 12 weeks

SECONDARY OUTCOMES:
Brief Pain Inventory - Pain severity | 12 weeks
Brief Pain Inventory - Pain interference | 12 weeks
Quantitative Sensory Testing - Vibration threshold | 12 weeks
Quantitative Sensory Testing - Electrical stimuli tolerance | 12 weeks
Numeric Pain Rating Scale - Back pain | 12 weeks